CLINICAL TRIAL: NCT00327548
Title: Treatment of Functional Abdominal Pain in Children:Evaluation of Relaxation/Guided Imagery and Chamomile Tea as Therapeutic Modalities
Brief Title: Use of Guided Imagery for Functional Abdominal Pain in Children:
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NIH 5P50-AT00008
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2006-10-05 (Estimated); Status verified 2002-07

CONDITIONS: Functional Abdominal Pain
MeSH Terms: interventions — Imagery, Psychotherapy

INTERVENTIONS:
Behavioral: guided imagery

SUMMARY:
The purpose of the study is to evaluate the effectiveness of relaxation, with or without guided imagery, for treating children with functional abdominal pain. The study will evaluate a child's ability to decrease the amount of pain with these techniques to allow continuation of normal daily activities at home and at school. The hypothesis is that these relaxation techniques will help decrease reports of abdominal pain and improve levels of activity.

ELIGIBILITY:
Inclusion Criteria:

at least 3 episodes of abdominal pain over the previous 3 months normal complete blood count, sedimentation rate, urinalysis stable on current medications English speaking -

Exclusion Criteria:

unwillingness to participate chronic gastrointestinal disease cognitive-developmental delay major dissociative disorder

-

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult

PRIMARY OUTCOMES:
Level of pain
number of days of pain
missed activities

CONTACTS AND LOCATIONS:
Overall Officials: Fayez K Ghishan, MD, Study Chair — University of Arizona